CLINICAL TRIAL: NCT04865276
Title: Adaptation and Evaluation of a Culturally and Gender Relevant Tobacco Cessation Among Women in Brazil: An Integrated mHealth Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007350
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Integrated tobacco cessation intervention delivered by Community Health Workers with the support of an App (mHealth) + Tobacco cessation program at the public health system
  Interventions: Behavioral: Integrated tobacco cessation intervention delivered by Community Health Workers with the support of an App (mHealth) + Tobacco cessation program at the public health system
- Control (Active Comparator): Home visit by a Community Health Worker during which the participant is scheduled to attend the tobacco cessation program at the public health system
  Interventions: Behavioral: Integrated tobacco cessation intervention delivered by Community Health Workers with the support of an App (mHealth) + Tobacco cessation program at the public health system

INTERVENTIONS:
Behavioral: Integrated tobacco cessation intervention delivered by Community Health Workers with the support of an App (mHealth) + Tobacco cessation program at the public health system — Integrated tobacco cessation intervention delivered by Community Health Workers with the support of an App (mHealth) + Tobacco cessation program at the public health system

SUMMARY:
We developed and established the efficacy of a theory-based, culturally- and gender-relevant Community Health Worker (CHW) intervention for low-income Brazilian women that augments the tobacco cessation program offered through the public health system. This study represents the continuation of our gender-relevant tobacco control efforts in Brazil by proposing the adaptation of this CHW-delivered tobacco cessation program to be integrated with mHealth support through mobile devices (App). We are proposing an integrated CHW-mHealth application that (a) is culturally- and gender-relevant, (b) is theory-based (Social Cognitive Theory), (c) considers the existing structure of the Brazilian health care system, and (d) will be adapted based on an efficacious intervention as well as salient features of other mHealth applications that have been shown to be successful in engaging users. During phase I we will make the adaptations and determine feasibility of a CHW-delivered intervention that is integrated with a mHealth tobacco cessation application (interactive App for participants and tracking system for CHWs) through formative assessments among all involved stakeholders, pretesting, and pilot testing of the intervention. In phase II we will assess the effectiveness of the integrated CHW-mHealth tobacco cessation intervention through a group randomized trial with towns as the unit of randomization (8 towns, N=344). The comparison group will be the same as the previous intervention (consisting of a home visit by a CHW during which the participant is scheduled to attend the tobacco cessation program at the neighborhood public health clinic) to allow for comparisons. We hypothesize that at 6-months, women smokers who receive the integrated CHW-mHealth intervention will have significantly higher 7-day point prevalence abstinence (defined as no cigarettes in the past 7 days) than women smokers in the control condition. Self-report will be verified through measurement of exhaled carbon monoxide levels among 30% of participants. If shown to be effective, this approach could be utilized as a model for a population-based intervention in low-resource settings, including rural and disadvantaged women in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Current tobacco use
* Willingness to quit tobacco use
* resident in the town assigned to intervention or control

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who self-identify as women
Enrollment: 431 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence (defined as no cigarettes in the past 7 days) | 6 months
  Nicotine abstinence as measured by self-report and CO

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No